CLINICAL TRIAL: NCT05715125
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of VTX958 in Patients With Active Psoriatic Arthritis
Brief Title: VTX958 Versus Placebo for the Treatment of Active Psoriatic Arthritis (Tranquility-PsA)
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: sponsor decision
Sponsor: Ventyx Biosciences, Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VTX958-203
Record Dates: First submitted 2023-01-19; First posted 2023-02-06 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Psoriatic Arthritis
Keywords: TYK2 inhibitor; Psoriatic arthritis; Ventyx; VTX958; Tranquility
MeSH Terms: conditions — Arthritis, Psoriatic

STUDY DESIGN:
Intervention Model Description: Participants are randomly assigned at the beginning of the study to either Dose A, Dose B, or placebo group, where they stay for the remainder of the study.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: The study has a double-blind design, meaning that the participant, care provider, and investigator will not know what treatment group each participant has been assigned to. This blinding will last from randomization until the end of the study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- VTX958 Dose A (Experimental)
  Interventions: Drug: Dose A VTX958
- VTX958 Dose B (Experimental)
  Interventions: Drug: Dose B VTX958

INTERVENTIONS:
Drug: Dose A VTX958 — Dose A VTX958
  Arms: VTX958 Dose A
Drug: Dose B VTX958 — Dose B VTX958
  Arms: VTX958 Dose B
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The objective of this study is to evaluate if VTX958 is safe and effective in adult participants with active Psoriatic Arthritis. Approximately 195 eligible participants will take VTX958 Dose A, VTX958 Dose B, or matching placebo (no active drug) for 16 weeks and then move on to a 36 week Long Term Extension (LTE). The study will include 16 weeks of treatment, 36 weeks of LTE, and a 30-day follow-up period.

DETAILED DESCRIPTION:
This is a Phase 2, multicenter, randomized, double-blind, placebo-controlled, parallel group study to evaluate the efficacy and safety of two doses of VTX958 tablets, Dose A and Dose B, in adults with active Psoriatic Arthritis. Approximately 195 participants will be assigned in a 1:1:1 ratio to one of three groups, VTX958 Dose A, VTX958 Dose B, or placebo, for 16 weeks and then move on to a 36 week Long Term Extension (LTE). The study consists of a 30-day screening period, a 16 week double-blind treatment period, 36 weeks of LTE, and a 30 day follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with Psoriatic Arthritis for 6 months or more prior to Screening
* Documented history or active signs of at least 1 confirmed lesion of plaque psoriasis and/or nail changes attributed to psoriasis
* Active PsA as defined by 3 or more swollen joints and 3 or more tender joints at Screening and Day 1
* Women must not be of childbearing potential or must agree to use a highly effective contraception during the study and for 30 days after the last dose of the study product
* Men with a partner who is of childbearing potential must agree to use condoms during the study and for 90 days after the last dose of study product

Exclusion Criteria:

* Has non-plaque psoriasis at Screening or Day 1
* Has inflammatory bowel disease or active uveitis
* Has a history of chronic or recurrent infectious disease
* Has a known immune deficiency or is immunocompromised
* Has hepatitis B or hepatitis C infection, human immunodeficiency virus (HIV), acquired immunodeficiency syndrome (AIDS), or active tuberculosis (TB) at screening

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 205 (Actual)
Dates: Start 2023-01-31 (Actual); Primary Completion 2024-01-02 (Actual); Study Completion 2024-01-02 (Actual)

PRIMARY OUTCOMES:
Proportion of participants achieving 20% improvement in American College of Rheumatology criteria (ACR20) at Week 16 | Week 16
  Number of participants reaching ACR20 at week 16, compared to the total number of participants in each cohort
Incidence of Treatment Emergent Adverse Events (TEAEs) from week 0 through week 16 | Week 16
  The number and proportion of participants who have at least 1 TEAE after exposure to the study drug

SECONDARY OUTCOMES:
Change from baseline in Health Assessment Questionnaire - Disability Index (HAQ-DI) scores at Week 16 | Week 16
  HAQ-DI assesses functional ability. It is a 20 question instrument that assesses the degree of difficulty with accomplishing tasks in 8 functional areas (dressing and grooming, arising, eating, walking, hygiene, reach, grip, and activities of daily living). Responses in each functional area are scored from 0 (no difficulty) to 3 (inability to perform a task in that area). The overall HAQ-DI score is the mean of the 8 functional area scores and ranges from 0 to 3. Lower scores are indicative of improved functional ability.
Proportion of participants achieving 75% reduction in the Psoriasis Area and Severity Index (PASI75) score at Week 16, in participants with at least 3% body surface area (BSA) involvement at baseline | Week 16
  PASI is used to assess the severity of psoriasis and response to therapy. Each body region is evaluated separately for body surface area percentage of involvement and translated to numeric score ranging from 0 (no involvement) to 6 (90 to 100% involvement) and for erythema, induration, and scaling, each is rated on scale of 0 to 4 (from none to maximum severity). PASI numeric scores range from 0 (no psoriasis) to 72 (maximal disease). Higher scores indicate more severe disease.
Change from baseline in Short Form Health Survey - 36 items (SF-36) physical component score (PCS) at Week 16 | Week 16
  SF-36 is a 36-item, patient-reported measure of health status and quality of life, which includes 8 domains (physical functioning, physical role functioning, bodily pain, general health perception, vitality, social functioning, emotional role functioning, and mental health). Each of the 8 domains contribute in different proportions to the physical component summary (PCS) score and the mental component summary (MCS) score, which are normalized to general US population norms and range from 0 to 100 (where higher scores correspond to a better quality of life).
Proportion of participants achieving 50% improvement in American College of Rheumatology criteria (ACR50) at Week 16 | Week 16
  Number of participants reaching ACR50 at week 16, compared to the total number of participants in each cohort
Proportion of participants achieving 70% improvement in American College of Rheumatology criteria (ACR70) at Week 16 | Week 16
  Number of participants reaching ACR70 at week 16, compared to the total number of participants in each cohort

CONTACTS AND LOCATIONS:
Overall Officials: Matt Cascino, MD, Study Director — Ventyx Biosciences, Inc
Locations (46):
- United States (15):
  - Site # 840001, Phoenix, Arizona
  - Site # 840016, Newport Beach, California
  - Site # 840004, Clearwater, Florida
  - Site # 840014, Miami Lakes, Florida
  - Site # 840017, Lexington, Kentucky
  - Site # 840018, Okemos, Michigan
  - Site #840012, Saint Clair Shores, Michigan
  - Site # 840019, Eagan, Minnesota
  - Site # 840003, Middleburg Heights, Ohio
  - Site # 840007, Duncansville, Pennsylvania
  - Site # 840010, Baytown, Texas
  - Site # 840006, Lubbock, Texas
  - Site # 840015, Mesquite, Texas
  - Site # 840011, Beckley, West Virginia
  - Site # 840008, South Charleston, West Virginia
- Bulgaria (3):
  - Site # 100004, Haskovo
  - Site # 100001, Plovdiv
  - Site # 100002, Plovdiv
- Czechia (5):
  - Site # 203004, Hlučín
  - Site # 203001, Ostrava
  - Site # 203003, Pardubice
  - Site # 203005, Prague
  - Site # 203002, Zlín
- Germany (2):
  - Site # 276002, Berlin
  - Site # 276001, Hamburg
- Hungary (3):
  - Site # 348003, Budapest
  - Site # 348001, Hódmezővásárhely
  - Site # 348004, Kistarcsa
- Poland (15):
  - Site # 616015, Gdynia
  - Site # 616007, Katowice
  - Site # 616010, Krakow
  - Site # 616009, Lodz
  - Site # 616012, Lodz
  - Site # 616014, Lodz
  - Site # 616013, Lublin
  - Site # 616002, Nadarzyn
  - Site # 616011, Olsztyn
  - Site # 616004, Poznan
  - Site # 616008, Torun
  - Site # 616006, Warsaw
  - Site #616001, Warsaw
  - Site # 616003, Wroclaw
  - Site # 616016, Wroclaw
- Spain (3):
  - Site # 724002, A Coruña
  - Site # 724005, Lleida
  - Site # 724001, Seville

IPD SHARING:
Plan to Share IPD: Undecided